CLINICAL TRIAL: NCT06669455
Title: SENSS (Stress, Exercise, Nutrition, Sleep, Self-management): an Integrated, Personalized and Stepped Care Lifestyle Approach for People with Parkinson's Disease: a Randomized Controlled Trial
Brief Title: An Integrated and Personalized Lifestyle Approach for People with Parkinson's Disease
Acronym: SENSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 115891
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Lifestyle; Personalized; Stepped Care; Quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group receiving:
  * Intake with lifestyle coach
  * Usual Care
  * Integrated, combined lifestyle approach (SENSS), including continuous monitoring by lifestyle coach.
  Interventions: Behavioral: Personalized and combined lifestyle approach
- Control (No Intervention): Control group receiving:
  * Intake with lifestyle coach
  * Usual care

INTERVENTIONS:
Behavioral: Personalized and combined lifestyle approach — In the SENSS approach five different and complementary lifestyle domains (self-management, exercise, nutrition, sleep and stress) are combined. The process will be guided by a lifestyle coach. The intervention is personalised for each participant. The personal goals are decided based on 'shared decision making' together with the lifestyle coach after using a Parkinson lifestyle decision aid. The level of guidance needed throughout the intervention is based on a 'stepped care approach'.
  Arms: Intervention

SUMMARY:
The goal of this study is to investigate the effects of a combined lifestyle program on the quality of life in people with Parkinson's Disease.

Participants will be randomly assigned to one of two groups, both receiving standard care, a Parkinson Lifestyle Decision aid and an intake meeting with a lifestyle coach. One group will work on their goals independently, while the other group will get guidance from the lifestyle coach throughout the 12-month program. The program focuses on self-management, exercise, nutrition, sleep and stress.

Participants will complete questionnaires after 0, 6 and 12 months, and use a wearable sensor for two weeks. The main outcome is quality of life over 12 months, measured with the PDQ-39 questionnaire. The study also examines personal goal achievements, symptom changes, and the economic effects of the program.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (idiopathic) in all stages of severity
* Proficient in Dutch, for both the data collection (questionnaires) and the intervention (all of the apps/modules are in Dutch)
* Aged 18 or older

Exclusion Criteria:

* Cognitive impairments that do not allow to fill out the questionnaires, as judged by the researcher during the screening call.
* Not in possession of or no access to an electronic device that allows for (video) calls with a lifestyle coach, and to complete questionnaires.
* Planned surgery or a planned major change in healthcare provision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life measured with the PDQ-39. | Measured at baseline, and after 6 and 12 months.
  The PDQ-39 consists of 39 questions across 8 dimensions of daily living including relationships, social situations and communication. Item scores range on a 5-point scale from "never" to "always". Both the total score of the PDQ-39 and the scores for each of the 8 dimensions are considered primary outcomes.

SECONDARY OUTCOMES:
Health related quality of life | Measured at baseline, and after 6 and 12 months.
  EuroQol 5D-5L (EQ-5D-5L); The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'.
Parkinson's Disease Symptoms | Measured at baseline, and after 6 and 12 months.
  The Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) part 1b and part 2. Questions are answered using a 0-4 likert scale ranging from 0 normal to 4 severe.
Fatigue | Measured at baseline, and after 6 and 12 months.
  Fatigue Severity Scale (FSS); This questionnaire consists of nine questions, each rated on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates greater fatigue or a more significant impact of fatigue on daily life.
Goal Attainment | Measured at baseline, and after 6 and 12 months.
  The visual analogue scale (VAS) is used to evaluate the lifestyle goals that participants set at the start of the intervention. The VAS is a non-specific measurement tool where patients rate their experience of a given sensation on a scale from 0 to 10.
Diet quality | Measured at baseline, and after 6 and 12 months.
  The Dutch Healthy Diet index 2015 (DHD15-index) consists of fifteen components representing the fifteen food-based Dutch dietary guidelines of 2015. Per component the score ranges between 0 and 10, resulting in a total score between 0 (no adherence) and 150 (complete adherence).
Mood (Anxiety and Depression) | Measured at baseline, and after 6 and 12 months.
  The Hospital Anxiety and Depression Scale (HADS) measures symptoms of anxiety and depression using a 14-item self-report questionnaire, over the past four weeks. It consists of a 7-item anxiety subscale and a 7-item depression subscale. Higher scores on the HADS indicate more symptoms, with a total score range of 0-42.
Physical activity level | Measured at baseline, and after 6 and 12 months.
  The LASA Physical Activity Questionnaire (LAPAQ) consists of 37 items designed to measure physical activities performed over the past week. The questionnaire assesses the frequency and duration of various physical activities. A higher score on the LAPAQ indicates a greater amount of time spent on physical activities.
Insomnia | Measured at baseline, and after 6 and 12 months.
  The Insomnia Severity Index (ISI) consists of seven items that assess various aspects of insomnia. The questionnaire includes the insomnia severity, satisfaction with sleep and impact on daily functioning. Each item is rated on a five-point Likert scale from 0 (not at all) to 4 (extremely), based on the last two weeks. The total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Sleepiness | Measured at baseline, and after 6 and 12 months.
  The Epsworth Sleepiness Scale (ESS) is a questionnaire that measures daytime sleepiness by assessing the likelihood of dozing or sleeping in eight different situations on a scale from 0 (would never doze or sleep) to 3 (high chance of dozing or sleeping). The total score ranges from 0 to 24, with higher scores indicating greater sleepiness.
Self-Efficacy | Measured at baseline, and after 6 and 12 months.
  The General Self-Efficacy Scale (GSES) is a 10-item questionnaire (total score range of 10-40) designed to measure a general sense of perceived self-efficacy. A higher score represents higher self-efficacy.
Ilness Acceptance | Measured at baseline, and after 6 and 12 months.
  Acceptance of Disease and Impairments Questionnaire (ADIQ); The questionnaire contains 14 items with a 4-point Likert scale ranging from 1 (disagree) to 4 (entirely agree).
Coping | At baseline.
  The ways of coping questionnaire (WCQ); Measures coping on eight dimensions. The questionnaire consists of 67 statements regarding coping in stressful situations. Participants have to score how much they think each statement applies to their situation on a 4-points Likert scale ranging from 0 ("does not apply and/or not used") to 3 ("used a great deal").
Self-management | Measured at baseline, and after 6 and 12 months.
  The Patient Activation Measure (PAM) is a 13-item survey that assesses an individual's self-reported knowledge, skills, and confidence in managing their health or chronic condition. Each item is rated on a 4-point Likert scale from "totally disagree" to "totally agree" or "non-applicable.
Change in physical activity from baseline to 12 months | Measured one week at baseline and one week after 12 months.
  Movement data captured with accelerometry data from a wrist worn wearable sensor (Empatica EmbracePlus).
Change in sleep time from baseline to 12 months | Measured one week at baseline and one week after 12 months.
  Captured with accelerometry and photoplethysmogry data from a wrist worn wearable sensor (Empatica EmbracePlus).
Change in sleep quality from baseline to 12 months | Measured one week at baseline and one week after 12 months.
  Captured with accelerometry and photoplethysmogry data from a wrist worn wearable sensor (Empatica EmbracePlus).

OTHER OUTCOMES:
Healthcare costs | At 6 and 12 months.
  Data on the used healthcare services used in the past 6 months will be collected with a questionnaire. The calculation uses tarrifs as determined for services for the healthcare in the Netherlands.
Intervention costs | During the intervention (from baseline until 12 months).
  The costs of the intervention consists of the amount of guidance provided by the lifestyle coach and the facilities used within the intervention, such as usage of a digital tool or online training. In the monitoring sessions with the lifestyle coach participants are asked what facilities they used in the prior period. This is registered by the lifestyle coach for each participant.
Process Evaluation | After completion of the 12 months intervention.
  In a process evaluation, caried out alongside the RCT, we aim to explore the experiences of participants and the lifestyle coaches with the SENSS approach. This process evaluation will take place through interviews with a selection of the participants and the lifestyle coaches.
Caregiver strain | Measured at baseline, and after 6 and 12 months.
  If the participants have a caregiver that is willing to participate in the study they receive a questionnaire and some follow-up questions about their task as caregiver and working life.
  Care Giver Strain Index (CSI); consists of 13 yes/no questions about the perceived strain. A higher score represents more strain.
  The caregivers will receive some questions about the amount of care they give and if/how this affects their working life. The results of these questions will be used in the analysis on (socio)economic impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands